CLINICAL TRIAL: NCT02223299
Title: A Randomized Double-Blind Placebo-Controlled Pilot Study of L-tyrosine and L-tryptophan in Depressed Patients Receiving L-methylfolate and and SSRI
Brief Title: Pilot Study: Combining Nutritional Supplements With Standard Antidepressant to Treat Depression.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never approved by the IRB and the PI left the VA
Sponsor: John D. Dingell VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 553Schanzer0002
Record Dates: First submitted 2014-08-19; First posted 2014-08-22 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Depression
Keywords: Depression; SSRI; Nutritional Supplements; Beck Depression Scale
MeSH Terms: conditions — Depression | interventions — Tyrosine; Tryptophan; 5-methyltetrahydrofolate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deplin w Supplements (Experimental): deplin 15mg plus L-Tyrosine 6g/d and L-Tryptophan 2g/d for 30 days
  Interventions: Dietary Supplement: L-tyrosine; Dietary Supplement: L-Tryptophan; Drug: deplin
- Deplin w placebo (Placebo Comparator): deplin 15mg daily plus Placebo A and Placebo B for 30 days
  Interventions: Drug: deplin; Other: Placebo A; Other: Placebo B

INTERVENTIONS:
Dietary Supplement: L-tyrosine — 6g/d daily for 30 days
  Arms: Deplin w Supplements
Dietary Supplement: L-Tryptophan — 2g/d daily for 30 days
  Arms: Deplin w Supplements
Drug: deplin — 15mg daily for 30 days
  Other Names: L-methylfolate
Other: Placebo A — a sugar-pill that looks like a real medication
  Arms: Deplin w placebo
Other: Placebo B — a sugar-pill that looks like a real medication
  Arms: Deplin w placebo

SUMMARY:
**This study never received IRB approval and no participants were ever enrolled** The purpose of this study is to determine if adding over the counter nutritional supplements will have a benefit to participants currently taking prescribed antidepressants who have not experienced complete remission of their depression symptoms.

DETAILED DESCRIPTION:
Inclusion Criteria:

Detroit VA Patients with major depression, mild to moderate treated with an SSRI and not having complete remission of symptoms as defined by "feeling their normal selves"

Randomized into two groups:

Experimental: will receive month supply of deplin 15mg, L-tyrosine 6g/d into 2 divided doses, and L-tryptophan 2g/d into 2 divided doses.

Control: will receive month supply of deplin 15mg , and 2 placebo pills.

Beck Depression Scale (BDI-2) to be administered at baseline and every 2 weeks for 1 month.

ELIGIBILITY:
**This study never received IRB approval and no participants were enrolled**

Inclusion Criteria:

* Veterans Administration Medical Center patients with major depression, mild to moderate treated with an SSRI and not having complete remission of symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Benefit of nutritional supplement | 30 days
  Through participant interviews and Beck Depression scale determine if adding nutritional supplements improve or resolve complete remission of depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- John D Dingell VA Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
This study never received IRB approval and never enrolled any participants. ClinicalTrials.gov entry should be removed.